CLINICAL TRIAL: NCT04120987
Title: The Incidence of Ocular Inflammation as Defined by the Inflammadry Assay in 250 Consecutive Cataract Patients and Their Response to Treatment With Xiidra
Brief Title: Ocular Inflammation in Cataract Patients and Response to Treatment With Xiidra
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Administrative
Sponsor: Bucci Laser Vision Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR-USA-002133
Record Dates: First submitted 2019-09-25; First posted 2019-10-09 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Dry Eye
Keywords: cataract; lifitegrast; dry eye syndrome; ocular surface inflammation; hyperosmolarity; MMP-9
MeSH Terms: conditions — Dry Eye Syndromes; Cataract | interventions — lifitegrast; Ophthalmic Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lifitegrast (Active Comparator): One drop of Lifitegrast Ophthalmic Solution 5% will be instilled into each eye twice daily (approximately 12 hours apart) using a single-use conainer.
  Interventions: Drug: Lifitegrast 5% Ophthalmic Solution
- Control (No Intervention): No treatment

INTERVENTIONS:
Drug: Lifitegrast 5% Ophthalmic Solution — BID OU
  Arms: Lifitegrast

SUMMARY:
To determine if the use of Xiidra® reduces ocular surface inflammation in preoperative and postoperative cataract patients.

DETAILED DESCRIPTION:
Single-center, prospective, randomized, investigator-initiated study

250 cataract patients, aged 60 or older, will be tested for ocular surface inflammation with the InflammaDry® immunoassay

Patients with bilateral positive MMP-9 will be randomized into a group treated with Xiidra two weeks preoperatively and six weeks postoperatively or a group not treated with Xiidra

The investigator hypothesizes that treatment with Xiidra prior to routine cataract surgery will significantly improve the quality of keratometry readings and BCVA.

ELIGIBILITY:
Inclusion Criteria:

* Positive for MMP-9 bilaterally as assessed by the Inflammadry assay

Exclusion Criteria:

* Negative Inflammadry assay in either eye
* Active diabetic retinopathy, uncontrolled glaucoma, uncontrolled uveitic inflammation
* Ocular surface diseases that might confound the interpretation of the InflammaDry assay

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2022-06-25 (Actual); Study Completion 2022-06-25 (Actual)

PRIMARY OUTCOMES:
Compare the conversion rates of bilateral positive MMP-9 to negative in pre-cataract and post-cataract patients receiving treatment with Xiidra versus no Xiidra | 12 weeks
  Compare the conversion rates of bilateral positive MMP-9 to negative in pre-cataract and post-cataract patients receiving treatment with Xiidra versus no Xiidra

CONTACTS AND LOCATIONS:
Overall Officials: Frank A Bucci, Jr., MD, Principal Investigator — Bucci Laser Vision
Locations (1):
- Bucci Laser Vision, Wilkes-Barre, Pennsylvania, United States